CLINICAL TRIAL: NCT02909660
Title: What Are You Looking for? Psychometric and Experimental Analyses of Reassurance Seeking in Obsessive-compulsive Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties / lack of participants
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Rachael Neal, Doctoral student, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30006114
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Support-seeking intervention (Experimental): Cognitive-behavioural therapy intervention that guides participants to seek support rather than reassurance; participants' significant others are asked to provide support rather than reassurance.
  Interventions: Other: Cognitive-behavioural therapy
- Family accommodation reduction intervention (Active Comparator): Cognitive-behavioural therapy intervention that guides participants' significant others to withhold reassurance when it is requested; participants are asked to refrain from seeking reassurance.
  Interventions: Other: Cognitive-behavioural therapy

INTERVENTIONS:
Other: Cognitive-behavioural therapy — Empirically-supported psychological intervention for various mental health concerns including obsessive-compulsive disorder (OCD). Includes components to foster cognitive (i.e., thinking) and behavioural changes.

SUMMARY:
This study evaluates the efficacy and acceptability of two cognitive-behavioural interventions for reassurance seeking behaviour in obsessive-compulsive disorder (OCD), a family accommodation reduction protocol vs. a novel support-seeking protocol. Half of participants will be randomly assigned to participate in the support-seeking intervention, whereas the other half will participate in the family accommodation reduction intervention.

DETAILED DESCRIPTION:
An existing family accommodation reduction intervention to reduce reassurance seeking behaviour in OCD (which represents treatment as usual, or TAU) is being compared to a novel support-seeking intervention to determine which is more efficacious and acceptable to participants.

The TAU protocol asks participants to make an agreement with their significant others to withhold reassurance when it is sought. It is believed that this behaviourally-based intervention encourages extinction of reassurance seeking over time by eliminating reinforcement of the behaviour by significant others.

The support-seeking intervention asks participants to move towards adaptively seeking support from a significant other to manage anxiety or distress rather than seeking reassurance. Significant others are taught to provide support rather than reassurance. It is believed that support-seeking may reduce reassurance seeking behaviour because it helps participants manage the anxiety or distress that underlies the requests for reassurance without interfering with disconfirmatory learning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD
* Engaging in reassurance seeking more than once a day about the same thing
* Willingness to allow the experimenter to contact a significant other from whom the participant seeks reassurance regularly
* Ability to read, write, and communicate in English

Exclusion Criteria:

* Current suicidal ideation/intent
* Current substance abuse
* Psychosis
* Diagnosis of bipolar disorder (I or II)
* If participants are on medication they must be on a stable dose (i.e., have maintained a consistent dose for at least three months) and agree not to change their medication regimen for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Self-reported reassurance seeking behaviour | 5 weeks (baseline through 3 week follow-up)
  Number of times participants self-report seeking reassurance per day
Self-reported support-seeking behaviour | 4 weeks (condition assignment through 3 week follow-up)
  Number of times participants in the support-seeking condition self-report seeking reassurance per day
Self-reported anxiety | 5 weeks (baseline monitoring through 3 week follow-up)
  Level of anxiety on average per day, self-rated from 0-100
One-week follow-up: Treatment Acceptability and Adherence Scale (TAAS; Milosevic, Levy, Alcolado, & Radomsky, 2015) | One-week follow-up
  Validated questionnaire assessing how acceptable participants find an intervention as well as ease of adherence.
One-week follow-up: Endorsement and Discomfort Scales (EDS; Tarrier, Liversidge, & Gregg, 2006) | One-week follow-up
  Validated questionnaire assessing acceptability of and discomfort caused by an intervention.
Three-week follow-up: Treatment Acceptability and Adherence Scale (TAAS; Milosevic, Levy, Alcolado, & Radomsky, 2015) | Three-week follow-up
  Validated questionnaire assessing how acceptable participants find an intervention as well as ease of adherence.
Three-week follow-up: Endorsement and Discomfort Scales (EDS; Tarrier, Liversidge, & Gregg, 2006) | Three-week follow-up
  Validated questionnaire assessing acceptability of and discomfort caused by an intervention.

SECONDARY OUTCOMES:
Change in self-reported reassurance-seeking | Baseline to one-week follow-up and baseline to three-week follow-up
  Pre-post assessment of change in the number of times per day that participants self-report reassurance seeking behaviour from the baseline monitoring week to the follow-up assessments.
Change in anxiety | Baseline (monitoring week 1) to end of reassurance provision week (monitoring week 2)
  Pre-post assessment of change in participants' self-reported anxiety ratings, as rated from 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No